CLINICAL TRIAL: NCT01481571
Title: Performance Study of New Media for Vitrification of Human Oocytes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitrolife (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Vitrolife-oocyte-vitri 01
Record Dates: First submitted 2011-11-18; First posted 2011-11-29 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-02

CONDITIONS: Infertility
Keywords: Media for vitrification/warming of human oocytes
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vitrification media and device (Experimental): Vitrification medium oocyte, warming medium oocyte and Rapid-i
  Interventions: Device: Vitrification medium oocyte, warming medium oocyte and Rapid-i

INTERVENTIONS:
Device: Vitrification medium oocyte, warming medium oocyte and Rapid-i — Media and device for vitrification of human oocytes

SUMMARY:
The purpose of this study is to evaluate safety and performance of Vitrolife´s new oocyte vitrification/warming media and the vitrification device Rapid-i™, when using vitrification as a cryopreservation method for human oocytes.

DETAILED DESCRIPTION:
A multi-center prospective sibling oocyte vitrification trial where, in the first phase, half of the patients' oocytes will be vitrified and warmed (experimental group). The remaining oocytes will not be vitrified and will serve as the control group. In the second phase all of the patients' oocytes will be vitrified and the embryo transfer will be performed in a following cycle. This simulates the situation of a normal cryopreservation embryo transfer. The study population consists of 20 women who will undergo a fresh IVF cycle during the study period. The primary objective in the first phase is to assess survival, fertilization and embryo development after oocyte vitrification/warming with the new media. The results will be compared with results from sibling oocytes which have not been vitrified. Secondary objectives are to assess the clinical results such as implantation, miscarriage and pregnancy rate as well as delivery rate and neonatal outcome.

The primary objective in the second phase is to assess the delivery rate after oocyte vitrification/warming with the new media. Secondary objectives are to assess survival, fertilization, embryo development, utilization rate, pregnancy rate and neonatal outcome on the previously vitrified and warmed oocytes. The results will be compared with results from a control group of patients, treated at the same clinics within the same time period, using the same inclusion and exclusion criteria. All patients who undergo embryo transfer will have a serum beta-hCG test conducted 14 days after oocyte retrieval. If positive, repeat beta-hCG testing will be conducted 2-4 days later. If appropriate, a pregnancy ultrasound will be conducted between 6-8 weeks gestation (menstrual age) to record gestational sac(s) and fetal heart beat. The delivery outcome will also be recorded. For patients with an unsuccessful treatment, there will be a follow-up period of 6 months after study completion. From this follow-up, data from frozen cycles, i.e. from embryos after oocyte vitrification, can be evaluated as well.

ELIGIBILITY:
Inclusion Criteria:

* Couple agreed to participate in study and has signed the Informed Consent Document before any study-related activities
* Patient age (female): 18-37 years (including oocyte donors)
* BMI 18-27 kg/m2 (female)
* 2 ovaries, normal uterine cavity (female)
* Day 3 FSH ≤ 10mIU, E2 <80 pg/mL and an AFC ≥12 (both ovaries, 3 mm or greater) (female)
* AMH >1 (female)
* Ejaculatory sperm (male)
* ICSI fertilization
* Long standard stimulation protocol
* English speaking

Exclusion Criteria:

* Previous participation in the study
* ≥2 previous failed IVF cycles
* Endometrioma
* Presence of a hydrosalpinx
* History of recurrent miscarriage (defined as ≥2 clinical recognized SABs)
* Not willing to have ICSI performed
* Cycle length >6 weeks [a diagnosis of PCOS will not exclude from the study unless typical cycle length is greater than 6 weeks; this criteria would exclude hypothalamic-hypogonadotropic patients]

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2012-01; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Embryo development after oocyte vitrification/warming. | 5 days after oocyte retrieval
  Embryo development, as number of good quality blastocysts, after oocyte vitrification and warming.

SECONDARY OUTCOMES:
Implantation rate of previously vitrified/warmed oocytes. | 4 weeks after embryo transfer
  Number of embryos implanted. Expressed as a percentage of number transferred.
Ongoing pregnancy rate | 3 months after embryo transfer
  Number of ongoing pregnancies at 3months. Expressed as a percentage of patients undergoing embryo transfer.
Live birth | 9 months after embryo transfer
  Number of lives births results from embryos transferred.

CONTACTS AND LOCATIONS:
Overall Officials: Marius Meintjes, Dr, Principal Investigator
Locations (2):
- United States (2):
  - The DFW Fertility Associates, Reproductive Endocrinology and Infertility, Dallas Fertility Centre, Dallas, Texas
  - Frisco IVF, Frisco, Texas